CLINICAL TRIAL: NCT03349268
Title: Pulsed UV Xenon Disinfection to Prevent Resistant Healthcare Associated Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Xenex Disinfection Services LLC (Industry); Detroit Medical Center (Other); Henry Ford Health System (Other); TEMPVA Research Group, Inc. (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, keith kaye, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01HS024709-01 (AHRQ)
Record Dates: First submitted 2017-11-02; First posted 2017-11-21 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Healthcare Associated Infection; Clostridium Difficile Infection; Infection Due to Multidrug Resistant Bacteria
MeSH Terms: conditions — Cross Infection; Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Two-armed crossover with an initial intervention period of 12 months, followed by a 6 month washout period and a second intervention period of 12 months. The 6 month washout period will be necessary because of the long-term survivability of eiHAIs, such as C. difficile, on environmental services.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All healthcare personnel (including device operators and environmental services staff) will be blinded to the intervention/sham status of the devices. In addition, the study personel including the PI and individuals performing data analysis, will be blinded to the intervention/sham status of the devices. The device status will be written on a piece of paper by the manufacturer with the serial numbers of each device indicated, sealed in an envelope and kept in a secure location by the study statistician for later retrieval when trial data analysis has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pulsed xenon ultraviolet light (PX-UV) Device Emitting Germicidal UV (Active Comparator): Pulsed xenon ultraviolet light (PX-UV) Device to be used to disinfect rooms following post-discharge terminal cleaning
  Interventions: Device: Pulsed xenon ultraviolet (PX-UV) Device; Device: Sham Device
- Sham Device - Non Emitting Germicidal UV (Sham Comparator): Sham Device to be run in rooms following post-discharge terminal cleaning. No Germicidal UV is emitted.
  Interventions: Device: Pulsed xenon ultraviolet (PX-UV) Device; Device: Sham Device

INTERVENTIONS:
Device: Pulsed xenon ultraviolet (PX-UV) Device — Two Detroit Medical Center (DMC) acute-care hospitals are being proposed for this project, Sinai-Grace Hospital (SGH) and Detroit Receiving Hospital (DRH). SGH is a 383-bed hospital, and DRH is a 248-bed hospital. The study will be conducted in eight hospital units in SGH and eight hospital units in DRH, including two medical intensive care units (ICUs), two surgical ICUs and 12 non-ICU medical-surgical wards. The 16 study units include a total of 379 beds.
  Devices will be deployed on these study units with the sham and intervention devices split evenly between SGH and DRH. Within each study site, the types of devices (PX-UV vs sham) will be assigned randomly to the units in Phase 1 and then switched in Phase 2.
Device: Sham Device — Two Detroit Medical Center (DMC) acute-care hospitals are being proposed for this project, Sinai-Grace Hospital (SGH) and Detroit Receiving Hospital (DRH). SGH is a 383-bed hospital, and DRH is a 248-bed hospital. The study will be conducted in eight hospital units in SGH and eight hospital units in DRH, including two medical intensive care units (ICUs), two surgical ICUs and 12 non-ICU medical-surgical wards. The 16 study units include a total of 379 beds.
  Devices will be deployed on these study units with the sham and intervention devices split evenly between SGH and DRH. Within each study site, the types of devices (PX-UV vs sham) will be assigned randomly to the units in Phase 1 and then switched in Phase 2.

SUMMARY:
The objective is to conduct a prospective, sham controlled, double-blinded, interventional crossover trial to compare standard terminal cleaning plus PX-UV (intervention) with standard terminal cleaning plus sham PX-UV (control) with crossover at 12 months, following a 6-month washout period. Outcome measures include the rates of HAIs, as well as the recurrence of genetically identical clinical strains of HAIs among patients on study units. The study will be conducted in 2 hospitals covering 16 total hospital units at Detroit Medical Center. Our central hypothesis is that the addition of PX-UV to standard terminal cleaning will be associated with a significant reduction in the rate of HAIs, as well as a reduction in the recovery of genetically identical strains of MDROs. The impact of PX-UV disinfection on rates of HAIs on study units will be determined by comparing rates of HAIs on a) study units where PX-UV is added to standard terminal cleaning practices to b) units where a sham UV disinfection system is added to standard terminal cleaning; and by comparing rates of HAIs on the same medical ward during each of two 12-month phases of a crossover study (one phase when a PX-UV device is added and one when a sham device is added to standard terminal cleaning).

The long-term goal of this project is to establish the efficacy of terminal cleaning plus PX-UV in reducing rates of HAIs due to the following multi-drug resistant organisms (MDROs): C. difficile, vancomycin-resistant enterococci (VRE), Klebsiella pneumoniae and Escherichia coli producing extended-spectrum beta-lactamases (ESBLs), methicillin-resistant Staphylococcus aureus (MRSA) and Acinetobacter baumannii.

At the conclusion of the proposed project, novel data will be generated from this rigorously controlled study regarding the effectiveness of PX-UV in reducing HAIs in a representative, real-world healthcare setting.

DETAILED DESCRIPTION:
In 2011, 721,800 healthcare-associated infections (HAIs) were reported in the United States. The hospital environment has been increasingly recognized as an important determinant of HAI acquisition and prevention of HAIs has become a top priority for the U.S. Department of Health and Human Services (HHS). Terminal cleaning of a patient room is recognized as a critically important process to help prevent HAIs and involves extensive cleaning and disinfection of the room after a patient has been discharged from the room and before the subsequent patient has been admitted to the room. Pulsed xenon ultraviolet light (PX-UV) has been shown to be effective in killing a variety of pathogens including endospores of Clostridium difficile. PX-UV works quickly - the entire cycle time for use in a hospital room is 15 minutes. To date, the clinical impact of adding PX-UV to terminal cleaning has not been demonstrated in clinical trials with sham controls or in a crossover design. The long-term goal of this project is to establish the efficacy of terminal cleaning plus PX-UV in reducing rates of HAIs due to the following multi-drug resistant organisms (MDROs): C. difficile, vancomycin-resistant enterococci (VRE), Klebsiella pneumoniae and Escherichia coli producing extended-spectrum beta-lactamases (ESBLs), methicillin-resistant Staphylococcus aureus (MRSA) and Acinetobacter baumannii. The objective of this application is to conduct a prospective, sham controlled, double-blinded, interventional crossover trial to compare standard terminal cleaning plus PX-UV (intervention) with standard terminal cleaning plus sham PX-UV (control) with crossover at 12 months, following a 6-month washout period. Outcome measures include the rates of HAIs, as well as the recurrence of genetically identical clinical strains of HAIs among patients on study units. The study will be conducted in 2 hospitals covering 16 total hospital units at Detroit Medical Center. Our central hypothesis is that the addition of PX-UV to standard terminal cleaning will be associated with a significant reduction in the rate of HAIs, as well as a reduction in the recovery of genetically identical strains of MDROs. The impact of PX-UV disinfection on rates of HAIs on study units will be determined by comparing rates of HAIs on a) study units where PX-UV is added to standard terminal cleaning practices to b) units where a sham UV disinfection system is added to standard terminal cleaning; and by comparing rates of HAIs on the same medical ward during each of two 12-month phases of a crossover study (one phase when a PX-UV device is added and one when a sham device is added to standard terminal cleaning). At the conclusion of the proposed project, novel data will be generated from this rigorously controlled study regarding the effectiveness of PX-UV in reducing HAIs in a representative, real-world healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the study units will be eligible
* Only patients who remain in the hospital for four calendar days or longer will be eligible for evaluation of eiHAI outcomes (the day of admission counts as calendar day one).
* Patients who do not develop an eiHAI at the time of unit discharge will be eligible for eiHAI outcomes for up to calendar 3 days following unit discharge.

Exclusion Criteria:

- All patients not cared for on study units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25732 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith S. Kaye, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhar S, Jinadatha C, Kilgore PE, Henig O, Divine GW, Todter EN, Coppin JD, Carter MJ, Chopra T, Egbert S, Carling PC, Kaye KS. Lowering the Acquisition of Multidrug-Resistant Organisms (MDROs) With Pulsed-xenon (LAMP) Study: A Cluster-Randomized, Controlled, Double-Blinded, Interventional Crossover Trial. Clin Infect Dis. 2024 Oct 15;79(4):1024-1030. doi: 10.1093/cid/ciae240. PMID 38743564

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PX-UV Disinfection, real or sham, occurred in rooms after each patient discharge when the room is unoccupied, so there is no direct risk to the patient from PX-UV disinfection treatments. Patients' medical treatment was not impacted in any way, and there was no additional testing in the study. The IRB waived consent. There is no numerical difference between started and complete, because definitionally, any patient in an included room was counted and their data was used to determine eiHAIs.
Groups:
- Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units: Pulsed xenon ultraviolet light (PX-UV) Device was used to disinfect rooms following post-discharge terminal cleaning: 2 Detroit Medical Center (DMC) acute-care hospitals were proposed for this project, Sinai-Grace Hospital (SGH) with 383 beds and Detroit Receiving Hospital (DRH) with 248; 8 hospital units in SGH and 8 hospital units in DRH, including 2 medical intensive care units (ICUs), 2 surgical ICUs and 12 non-ICU medical-surgical wards.
  Devices were deployed on these study units with the sham and intervention devices split evenly within SGH and DRH. Within each study site, the types of devices (PX-UV vs sham) were assigned randomly to the units in Phase 1 and then switched in Phase 2.
- Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units: Sham Device was run in rooms following post-discharge terminal cleaning. No Germicidal UV was emitted. 2 Detroit Medical Center (DMC) acute-care hospitals were proposed for this project, Sinai-Grace Hospital (SGH) with 383 beds and Detroit Receiving Hospital (DRH) with 248; 8 hospital units in SGH and 8 hospital units in DRH, including 2 medical intensive care units (ICUs), 2 surgical ICUs and 12 non-ICU medical-surgical wards.
  Devices were deployed on these study units with the sham and intervention devices split evenly between SGH and DRH. Within each study site, the types of devices (PX-UV vs sham) were assigned randomly to the units in Phase 1 and then switched in Phase 2.
- Patients Cared for on Both PX-UV and Sham Units: Despite the original study design where crossover occurred at the unit level, some patients were cared for on both a PX-UV unit as well as a Sham unit. The degree to which this occurred was unexpected, yet unavoidable. As a results, they are assigned to this arm to explain their exclusion from each of the single treatment arms. It was not part of the original intention of the study to evaluate patients who were in both study environments.
  Because these patients were exposed to both study environments, their outcomes could not be attributed to either study intervention.
Period: Overall Study
Arm/Group | Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units | Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units | Patients Cared for on Both PX-UV and Sham Units
Started | 9117 | 10296 | 6319
Completed | 9117 | 10296 | 6319
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Cared for on Both PX-UV and Sham Units: Despite the original study design where crossover occurred at the unit level, some patients were cared for on both a PX-UV unit as well as a Sham unit. The degree to which this occurred was unexpected, yet unavoidable.
- Total: Total of all reporting groups
Arm/Group | Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units | Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units | Patients Cared for on Both PX-UV and Sham Units | Total
Number analyzed (Participants) | 9117 | 10296 | 6319 | 25732
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (18.23) | 57.46 (18.41) | 61.50 (16.51) | 58.43 (17.98)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4253 | 4962 | 3018 | 12233
  Male | 4858 | 5333 | 3291 | 13482
  Unknown | 6 | 1 | 10 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 32 | 34 | 20 | 86
  Asian/Pacific Islander | 31 | 22 | 13 | 66
  Black or African American | 7142 | 8085 | 5212 | 20439
  White | 933 | 1025 | 419 | 2377
  Unknown/Not Reported/Other | 979 | 1130 | 655 | 2764
Region of Enrollment [Number; unit: participants]
  United States | 9117 | 10296 | 6319 | 25732

OUTCOME MEASURES:

1. Primary Outcome: Number of Environmentally-implicated Healthcare-Associated Infections (eiHAIs) Associated With the Additional Use of a PX-UV Disinfection Compared to Standard Terminal Cleaning
Description: PX-UV Device was used following each discharge on study units, with intervention devices emitting germicidal UV on 50% of the units and sham devices not emitting germicidal UV on 50% of the units.
Time Frame: 24 months (Two 12 month phases)
Population: It was not part of the original intention of the study to evaluate patients who were in both study environments.
  Because these patients were exposed to both study environments, their outcomes could not be attributed to either study intervention. Therefore the de facto "third arm" which accounts for them is not included in this analysis.
Measure: Number; unit: eiHAIs
Units Other Than Participants: patient days
Arm/Group | Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units | Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units
Number analyzed (Participants) | 9117 | 10296
Number analyzed (patient days) | 86800 | 94154
eiHAIs | 303 | 298
Statistical Analysis 1: Comparison: Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units vs Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units; Test type: Superiority; p = 0.23, Poisson regression

ADVERSE EVENTS:
Description: This is not a treatment trial. The PX-UV Disinfection, whether real or sham, occurred only in rooms following each patient discharge when the room was unoccupied, so there was no direct risk to the patient from PX-UV or sham disinfection treatments. Patients' medical treatment was not impacted in any way by this study, and they did not undergo any additional testing as part of the study. Therefore no AE data was collected or recorded.
Groups:
- Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units: Sham Device was run in rooms following post-discharge terminal cleaning. No Germicidal UV was emitted. 2 Detroit Medical Center (DMC) acute-care hospitals were proposed for this project, Sinai-Grace Hospital (SGH) with 383 beds and Detroit Receiving Hospital (DRH) with 248; 8 hospital units in SGH and 8 hospital units in DRH, including 2 medical intensive care units (ICUs), 2 surgical ICUs and 12 non-ICU medical-surgical wards.
Arm/Group | Patients Only on Pulsed Xenon Ultraviolet Light (PX-UV) Device Emitting Germicidal UV Units | Patients Cared for on Only Sham Device - Non Emitting Germicidal UV Units | Patients Cared for on Both PX-UV and Sham Units
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03349268/Prot_SAP_000.pdf